CLINICAL TRIAL: NCT02592759
Title: Effects of Upper Extremity Rehabilitation Using Smart Glove in Stroke
Brief Title: Effects of Upper Extremity Rehabilitation Using Smart Glove in Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was prematurely terminated due to slow recruitment.
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Shi-Uk Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-2015-74
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smart Glove Group (Experimental): The subjects will be treated with conventional occupational therapy for 30 minutes and smart glove treatment for 30 minutes. 5 treatments per week will be conducted a total of 2 weeks.
  Interventions: Device: Smart Glove Treatment
- Homework group (No Intervention): The subjects will be treated with conventional occupational therapy for 30 minutes and upper extremity rehabilitation homework which means the self training at bedside, for 30 minutes. 5 treatments per week will be conducted a total of 2 weeks.

INTERVENTIONS:
Device: Smart Glove Treatment — Smart glove is digital motion-based treatment device for stroke rehabilitation. The stroke patients wear this glove and hand motion is displayed on the computer monitor. They play games with this glove and are motivated to rehabilitation treatment because of fun.
  Arms: Smart Glove Group

SUMMARY:
The purpose of this study is to evaluate the therapeutic effects of smart glove which is motion-based program designed for upper extremity rehabilitation after stroke.

DETAILED DESCRIPTION:
This study will evaluate the therapeutic effects (upper extremity power, function and activity of daily living) of smart glove which is motion-based rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* CT or MRI proved 1st stroke patients with unilateral hemiplegia caused by stroke (ischemic, hemorrhagic, intracranial hemorrhage)
* 72 hours ~ 3 months after stroke
* Upper extremity hemiplegia with Brunnström stage 2-5.
* The patients can sit to receive treatment for at least 1 hour

Exclusion Criteria:

* The patients cannot perform occupational treatments because of severe hemineglect or hemianopia
* Contracture due to severe limitation of motion
* Upper extremity spasticity in the wrist and fingers with modified Ashworth scale > 2 points
* Fugl-Meyer Assessment-Wrist & Hand score >= 21 points
* moderate to severe cognitive dysfunction < MMSE 18 points
* Severe aphasia
* The patients who has been diagnosed as malignant tumor

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity change | Change from baseline points at 2 weeks and 6 weeks
  Evaluation tool for upper extremity function

SECONDARY OUTCOMES:
Brunnström stage change | Change from baseline stage at 2 weeks and 6 weeks
  Evaluation tool for recovery
Modified Barthel Index change | Change from baseline points at 2 weeks and 6 weeks
  Evaluation tool for the level of active daily living
Care Burden Scale change | Change from baseline points at 2 weeks and 6 weeks
  Evaluation tool to measure the care burden
Hand power change | Change from baseline power at 2 weeks and 6 weeks
  Hand power using hand-held dynamometer
Jebsen Hand function Test change | Change from baseline points at 2 weeks and 6 weeks
  Evaluation tool for upper extremity function
Box and Block Test change | Change from baseline points at 2 weeks and 6 weeks
  Evaluation tool for upper extremity function

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Uk Lee, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang MG, Yun SJ, Lee SY, Oh BM, Lee HH, Lee SU, Seo HG. Effects of Upper-Extremity Rehabilitation Using Smart Glove in Patients With Subacute Stroke: Results of a Prematurely Terminated Multicenter Randomized Controlled Trial. Front Neurol. 2020 Nov 9;11:580393. doi: 10.3389/fneur.2020.580393. eCollection 2020. PMID 33240205